CLINICAL TRIAL: NCT06094062
Title: Smartphone App-assisted Discontinuation of Short-term PPI Treatment - an Feasibility Study
Brief Title: Smartphone App-assisted PPI
Acronym: PIPPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-00588
Record Dates: First submitted 2023-09-27; First posted 2023-10-23 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-12

CONDITIONS: Heartburn; Dyspepsia
Keywords: Medication Adherence; Short-term Therapy; Proton Pump Inhibitors; Mobile Health; Implementation
MeSH Terms: conditions — Heartburn; Dyspepsia; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental)
  Interventions: Other: App-based treatment support

INTERVENTIONS:
Other: App-based treatment support — The intervention includes a smartphone app that patients will download on their smartphones. Medication intake, symptom course and well-being will be tracked over treatment duration. If symptoms worsen, the pharmacist will contact the patients and counsel them based on their adherence and well-being data. Patients who still have symptoms after the 30 days of treatment will receive a final counseling by the pharmacy, and if necessary will be forwarded to the treating physician.

SUMMARY:
Proton pump inhibitors (PPIs) are frequently prescribed for 30 days but taken infinitely. PPIs belong to the most often inappropriate medicines (PIMs). Correct intake of medicines (named adherence) can be supported by digital devices such as smartphone applications. The goal of this interventional study is to test the feasibility of an app-based treatment support provided by community pharmacists in patients prescribed a short-term PPI (30 days). The intervention consists in tracking medication intake, symptom course and well-being over the treatment duration of 30 days with the mednet app on patients' personal smartphones.

DETAILED DESCRIPTION:
This is an exploratory study in a primary care setting with community pharmacists recruiting patients who are newly prescribed a PPI for a short-term treatment (30 days). There is no control group and no randomization. After informed consent and installing the app on their personal smartphones, patients will answer three questions from the app once daily. The questions address medication intake (yes/no), symptom course (better, worse, identical, no symptoms) and well-being (satisfactory/needs improvement). Worsening of symptoms will trigger an alarm (via email) at the pharmacy. The pharmacist will call the patients and use information from adherence and well-being to consolidate a supporting counseling.

Feasibility and a frequency estimation of the interventions will be the focus of the study in view of a larger implementation study with community pharmacies. Further implementation outcomes will be assessed through interviews and surveys (satisfaction, interprofessional work).

ELIGIBILITY:
Inclusion Criteria:

* is ≥18 years old;
* has symptoms that suggest or correspond to gastroesophageal reflux disease (GERD);
* is newly prescribed a short-term PPI treatment;
* accepts to use of the smartphone app mednet during the study period;
* signs the informed consent form;
* understands and speaks (Swiss) German.

Exclusion Criteria:

* in the opinion of the pharmacist or physician, unlikely to comply with the study schedule or are unsuitable for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Patients with PPI treatment over 30 days | 30 days (treatment duration)
  Number of patients who started and stopped a PPI after 30 days

SECONDARY OUTCOMES:
Treatment extensions | 30 days (treatment duration)
  Number of PPI treatment extensions including reasons and number of additional days
Physicians' and pharmacists' satisfaction with the service | 2 weeks after study completion
  Physicians' and pharmacists satisfaction with the service including adherence report assessed through semi-structured interviews
Patients' satisfaction with the service | 2 weeks after the end of treatment
  Patients' satisfaction with the service including the app assessed through semi-structured interviews
Reliable diagnosis after PPI treatment | After 30 days (treatment duration)
  Number of reliable diagnosis after short-term PPI treatment including treatment extensions

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Arnet, Dr. PD, Principal Investigator — University of Basel, Pharmaceutical Care Research Group
Locations (2):
- Switzerland (2):
  - Goldene Engel Apotheke, Basel, Canton of Basel-City
  - TopPharm Apotheke am Spalebärg, Basel, Canton of Basel-City